CLINICAL TRIAL: NCT00268931
Title: Enhanced Developmental Training Experiences in Babies Born Preterm
Brief Title: Development Training in Babies Born Preterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24098
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Premature Birth
Keywords: premature birth; motor skills; learning; reaching
MeSH Terms: conditions — Premature Birth | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- True Control (No Intervention): This group is being enrolled as a true control group. This group will not participate in the movement training or social training however, they will be evaluated in the same way.
- Social Training (Experimental): This group underwent specific social interactions two times each day with their parents.
  Interventions: Behavioral: Social Training
- Movement Training (Experimental): This group of preterm infants underwent movement training two times per day with their parents.
  Interventions: Behavioral: Movement Training

INTERVENTIONS:
Behavioral: Movement Training — This group of infants underwent specific movement training activities two times per day with their parents.
  Arms: Movement Training
Behavioral: Social Training — This group underwent special social interactions with their parents two times each day.
  Arms: Social Training

SUMMARY:
The specific purpose of this study is to determine the effect of movement training on the onset of motor skills in babies born prematurely. We hypothesize that infants who participate in movement training will show advances in motor skills, visual attention, and toy-oriented behavior.

DETAILED DESCRIPTION:
The long term goal of this research program is to develop detailed intervention options for physical therapy treatment of very young preterm infants at risk for disability. The ability of infants to start reaching marks the beginning of an infants' ability to independently explore objects, and impacts development across multiple domains, including cognitive, language, and social. The aim of this study is to determine if bi-daily movement training will advance the reaching abilities of infants born preterm as compared to non-movement trained controls.

Movement Training Group:

Parents/Caregivers will be instructed to improve their infants' awareness and ability to reach for toys with their arms and legs by performing two sets of 10 minutes of daily exercises with them. The first 10 minutes will focus on improving awareness of their arms and toys (such as bells on their wrists). The second 10 minutes of activity that focuses on introducing infants to a task-space they rarely experience at this age, the task-space required for midline reaching (such as moving the infant's arm to a midline toy). An experimenter will visit each family in their homes every other week (the week that is not a testing week) to assure correctness of training, encourage full participation and answer any questions.

Social Training Group:

To control for increased social interaction that accompanies the enhanced training, parents of infants in this group will serve as a control group. Parent/Caregivers will be asked to perform 2x a day of 10 minutes face-to-face social interaction with their infants. Parents and infants will receive a 10 minute audio tape of popular kids' songs. They will be instructed to place infants supine or in a bouncy seat and interact with the infant visually and verbally during this time period along with the music.

After the study is completed, each group will be offered the training booklet that the opposite group received.

ELIGIBILITY:
Inclusion Criteria:

* Infants born less than 33 weeks gestation (up to and including 32 6/7 weeks)
* Infants born weighing less than 2500 grams

Exclusion Criteria:

* Orthopedic, visual or hearing impairments
* Fetal drug exposure

Ages: 6 Weeks to 11 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2004-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to evaluate the effectiveness of movement training in preterm babies. This will be measured by number of toy contacts, hand/foot-toy distance, duration of toy contact, and duration of visual attention. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jill C. Heathcock, MPT, Principal Investigator — University of Delaware; James C Galloway, Ph.D., Principal Investigator — University of Delaware
Locations (1):
- Christiana Care Health Systems, Newark, Delaware, United States

REFERENCES:
- [Background] Fagen JW, Morrongiello BA, Rovee-Collier C, Gekoski MJ. Expectancies and memory retrieval in three-month-old infants. Child Dev. 1984 Jun;55(3):936-43. PMID 6734328
- [Background] Heathcock JC, Bhat AN, Lobo MA, Galloway JC. The relative kicking frequency of infants born full-term and preterm during learning and short-term and long-term memory periods of the mobile paradigm. Phys Ther. 2005 Jan;85(1):8-18. PMID 15623358
- [Background] Heathcock JC, Bhat AN, Lobo MA, Galloway JC. The performance of infants born preterm and full-term in the mobile paradigm: learning and memory. Phys Ther. 2004 Sep;84(9):808-21. PMID 15330694
- [Background] Cherkes-Julkowski M. Learning disability, attention-deficit disorder, and language impairment as outcomes of prematurity: a longitudinal descriptive study. J Learn Disabil. 1998 May-Jun;31(3):294-306. doi: 10.1177/002221949803100309. PMID 9599962
- [Background] de Vries AM, de Groot L. Transient dystonias revisited: a comparative study of preterm and term children at 2 1/2 years of age. Dev Med Child Neurol. 2002 Jun;44(6):415-21. doi: 10.1017/s0012162201002298. PMID 12088310
- [Background] Angulo-Kinzler RM, Ulrich B, Thelen E. Three-month-old infants can select specific leg motor solutions. Motor Control. 2002 Jan;6(1):52-68. doi: 10.1123/mcj.6.1.52. PMID 11842270
- See also: University news article — http://www.udel.edu/PR/UDaily/2004/infant032604.html